CLINICAL TRIAL: NCT01152411
Title: Use of Autologous Bone Marrow Stem Cell Transplantation in the Treatment of Chronic Renal Failure in 5 Indian Patients - ABMST-CRF Study (Autologous Bone Marrow Stem Cell Transplantation-CRF)
Brief Title: Safety and Efficacy of Autologous Bone Marrow Stem Cells for Treating Chronic Renal Failure
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: International Stemcell Services Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISSL-AuBM-CRF
Record Dates: First submitted 2010-06-26; First posted 2010-06-29 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Renal Failure
Keywords: Renal Failure; Chronic Kidney Disease; Chronic Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous bone marrow stem cells (Experimental)
  Interventions: Other: Autologous bone marrow stem cells

INTERVENTIONS:
Other: Autologous bone marrow stem cells — Bone marrow stem cells; Single dose; Interventional fluoroscopy-guided injection into the renal artery.

SUMMARY:
Chronic renal failure (CRF, or "chronic kidney failure", CKF, or "chronic kidney disease", CKD) is a slowly progressive loss of renal function over a period of months or years and defined as an abnormally low glomerular filtration rate, which is usually determined indirectly by the creatinine level in blood serum.

CRF that leads to severe illness and requires some form of renal replacement therapy(such as dialysis) is called end-stage renal disease (ESRD). While renal replacement therapies can maintain patients indefinitely and prolong life, the quality of life is severely affected. Renal transplantation increases the survival of patients with stage 5 CKD significantly when compared to other therapeutic options; however, it is associated with an increased short-term mortality (due to complications of the surgery).

In view of the above, there is definitely an urgent need for finding different methods of treatment for these patients who cannot undergo established modalities of treatment or these have been tried unsuccessfully hence the inadequacy of current treatment modalities and insufficiency of donor organs for transplantation have driven a search for improved methods of dealing with renal failure. The rising concept of cell-based therapeutics has provided a framework around which new approaches are being generated, and its combination with advances in stem cell research stands to bring both fields to clinical fruition. Since CRF affects a large number of these patients who will lose their productive life, stem cell implantation can offer some promise of improved health.

In our present study, we want to evaluate the safety and efficacy (to know / observe for Proof of concept in five indian patients) if any, of autologous bone marrow derived stem cells injected into the Renal Artery in five (initially five patients, can be increased to ten patients after observing the initial results) patients with Chronic Renal Failure.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to give voluntary written (patients may not be able to write) consent.
2. Must be able to understand study information provided to him.
3. CKD patients of stage IV and ESRD with age 18 to 65 years.
4. Patient should be afebrile 24 hours prior to procedure.

Exclusion Criteria:

* Women who are pregnant or lactating
* Acute Renal Failure
* Severe co-morbidities like cardiac insufficiency, congestive cardiac failure, malignancy, infection, sepsis and bed sores.
* Haemoglobin level below 8g %
* Chronic kidney disease due to autoimmune aetiology, connective tissue disease, amyloidosis and storage disorders.
* Known bleeding or coagulation disorder.
* Known hematologic disease
* Poorly controlled hypertension
* Evidence of active malignancy within one year prior to randomization.
* Severe skin infection or osteomyelitis - the site of bone marrow aspiration potentially limiting the procedure.
* Have a known allergy to iodinated contrast
* Positive test results for HIV and AIDS complex, HCV, HbsAg and Syphilis.
* History of drug or alcohol abuse
* Patients on immunosuppressive therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2010-02; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Significant clinical improvement in serum creatinine and urine output (improvement in measured GFR by 50%) | 1 year
Number of patients reporting adverse effects as a measure of safety and tolerability | 1 year

SECONDARY OUTCOMES:
Improvement in renal biopsy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Balakrishna S, M.B.B.S, Study Director — International Stemcell Services Limited
Locations (1):
- St. Theresa's Hospital, Bengaluru, Karnataka, India